CLINICAL TRIAL: NCT01728467
Title: Phase 2 Randomised, Double-blind, Placebo-controlled, Cross-over Study for the Assessment of Glucose Metabolism Changes With RVX000222 in Individuals With Pre-diabetes
Brief Title: The Effects of RVX000222 on Glucose Metabolism in Individuals With Pre-diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Collaborators: Baker Heart and Diabetes Institute (Other); Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVX222-CS-010; Alfred Study No. 409/12 (Other: Baker IDI Heart and Diabetes Institute)
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — apabetalone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RVX000222, 200 mg daily (Experimental)
  Interventions: Drug: RVX000222
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo, RVX000222

INTERVENTIONS:
Drug: RVX000222 — capsule, 200 mg, administer with food, 100 mg twice daily 10-12 hrs apart, 31-35 days
  Other Names: RVX-208
  Arms: RVX000222, 200 mg daily
Drug: Placebo, RVX000222 — capsule, administer with food, twice daily 10-12 hrs apart, 31-35 days
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study builds on data that high-density lipoprotein (HDL) has a number of potentially beneficial effects including directly modulating glucose metabolism through multiple mechanisms. The primary objective of this study is to determine the effects of RVX000222 on postprandial plasma glucose in male individuals with impaired fasting glucose (IFG) or impaired glucose tolerance (IGT), during a frequently sampled oral glucose tolerance test (OGTT).

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-70 years, inclusive
* Body mass index (BMI): 25-40 kg/m2
* HDL cholesterol plasma levels: ≤1.4 mmol/L
* Pre-diabetes: Either impaired fasting glucose (IFG; 6.1-6.9mmol/L) or impaired glucose tolerance (IGT; 2 hour OGTT glucose 7.8-11.0mmol/L, WHO classification) as measured at Visit 1
* No current use or need for prescription or over-the-counter medication within four days of Visit 1
* Have given signed informed consent to participate in the study

Exclusion Criteria:

* Identification of any other medical condition requiring immediate therapeutic intervention
* Has received any over-the-counter medication including vitamins, herbal, or dietary supplements within four days of Visit 1 unless prior approval from the Investigator
* Tobacco use within six months of Visit 1 (including cigarettes, pipes, chewing tobacco)
* Elective surgery requiring general anaesthesia during the course of the study
* Clinically significant heart disease at Visit 1
* Clinically significant abnormal ECG at Visit 1
* Evidence of renal impairment defined as serum creatinine >1.5 mg/dL (133 μmol/L) or creatinine clearance of <60 mL/min
* History of hypertension or supine SBP >160mmHg or DBP >95mmHg as measured at Visit 1
* Evidence of type 2 diabetes (fasting plasma glucose ≥7.0mmol/L; 2 hour OGTT glucose ≥11.1mmol/L)
* Evidence of liver disease defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT) or total bilirubin >1.5 x upper limit of normal (ULN) at Visit 1
* History of malignancy within past 5 years
* History or evidence of drug or alcohol abuse within 12 months of Visit 1
* Use of other investigational drugs and/or devices at the time of enrolment, or within 30 days of Visit 1
* History of non-compliance to medical regimens or unwillingness to comply with the study protocol
* Any condition that in the opinion of the Investigators would confound the evaluation and interpretation of the data
* Persons directly involved in the execution of the protocol

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose following treatment with RVX000222 compared to placebo | 29-33 days
  The change in postprandial plasma glucose, defined as area under the glucose curve (AUGC) during a frequently sampled OGTT following RVX000222 treatment for 29-33 days as compared to placebo.

SECONDARY OUTCOMES:
Change in insulin secretion and insulin sensitivity following treatment with RVX000222 compared to placebo | 29-33 days
  The change in indices of insulin secretion (β-cell function) and insulin sensitivity during a frequently sampled OGTT following RVX000222 treatment for 29-33 days as compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Bronwyn Kingwell, Principal Investigator — Baker Heart and Diabetes Institute; Dr. Stephen Duffy, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker IDI Heart and Diabetes Institute 75 Commercial Road,, Melbourne, Victoria, Australia